CLINICAL TRIAL: NCT06752889
Title: Clinical and Radiographic Evaluation of Zinc Oxide Modified 3Mixtatin Versus Zical Root Canal Sealer in Root Canal Treatment of Necrotic Primary Molars.(A Randomized Clinical Trial and in Vitro Study)
Brief Title: Clinical and Radiographic Evaluation of Zinc Oxide Modified 3Mixtatin Versus Zical in Root Canal Treatment of Necrotic Primary Molars.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PED21-9
Record Dates: First submitted 2024-03-29; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-03

CONDITIONS: Necrotic Pulp; Primary Teeth
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group( 1): Control Group (pulpectomy using zic oxide eugenol based sealer Zical): (Active Comparator): Local anesthesia administration and rubber dam isolation will be carried out Access cavity will be prepared, necrotic pulp tissue will be removed using a sterile sharp spoon excavator.
  Cleaning and shaping of the root canals will be carried out using H files and continuous irrigation.
  Canal irrigation with 2.5% sodium hypochlorite will be carried out throughout the procedure.
  Sterile paper points will be used to dry the root canals. Zinc oxide eugenol based sealer (Zical) will be mixed into a thick paste and packed into the pulp chamber to fill the canal. (Chen& Zhong., 2017; Pramila., 2015) The access opening will be sealed with a glass ionomer cement , and the tooth will be restored with a stainless steel crown.
  Interventions: Other: Group( 1): Control Group (pulpectomy using zic oxide eugenol based sealer Zical):
- Group ( 2) Experimental group modified 3-MIX-TATIN): (Experimental): dified 3Mix-tatin will be prepared by mixing three commercially available antibiotics with simvastatin. After removing the coating materials, 3 types of antibiotics are pulverized by porcelain mortars and pestles to achieve fine powders. A total of 100 mg ciprofloxacin, 100 mg metronidazole, and 100 mg cefixime will be mixed in a ratio of 1: 1: 1. Two milligrams of simvastatin will be added to the drugs blend to form 3-Mix-tatin. Preparation of 3Mix-tatin will be trained and supervised by an expert pharmacist. 3Mixtatin will be stored in a tightly capped porcelain container, adding of silica gel in a bag inside the container to maintain low humidity. This powder will be mixed with zinc oxide eugenol based sealer called Zical which will act as a carrier or vehicle to form a creamy paste of 3Mixtatin at the time of application (Aminabadi et al., 2015; carvalho., 2016).
  Interventions: Other: Group ( 2) Experimental group modified 3-MIX-TATIN):

INTERVENTIONS:
Other: Group( 1): Control Group (pulpectomy using zic oxide eugenol based sealer Zical): — Zinc oxide eugenol based sealer (Zical) will be mixed into a thick paste and packed into the pulp chamber to fill the canal.
  Arms: Group( 1): Control Group (pulpectomy using zic oxide eugenol based sealer Zical):
Other: Group ( 2) Experimental group modified 3-MIX-TATIN): — Modified 3Mix-tatin will be prepared by mixing three commercially available antibiotics with simvastatin. This powder will be mixed with zinc oxide eugenol based sealer called Zical which will act as a carrier or vehicle to form a creamy paste of 3Mixtatin at the time of application
  Arms: Group ( 2) Experimental group modified 3-MIX-TATIN):

SUMMARY:
Primary molars with necrotic pulp or abscess are common unfortunate event faced in pediatric dentistry .The traditional treatment is either pulpectomy or extraction. ٍuccess of pulpectomy treatment is about 85% in abscessed primary teeth.

The aim of pulpectomy is to preserve teeth in a symptom free state until they are replaced by their successor naturally during the transition from primary to permanent dentition, thus avoiding extraction. The adequate restoration of the involved teeth may preserve the arch length reestablish the masticatory function and esthetics and prevent harmful tongue habits and speech alterations due to anterior teeth decay.

DETAILED DESCRIPTION:
The techniques available for management of necrotic primary molars are either pulpectomy or extraction, but according to guidelines American Academy of Pediatric Dentistry, extraction and space maintainer is a viable option but a successfully restored tooth is far superior space maintainer than an appliance. So preservation of primary molars is not only important for masticatory function but also for preservation of developing occlusion.

The rationale includes the chemical and mechanical removal of irreversibly inflamed or necrotic radicular pulp tissue, followed by root canal filling with a material that can resorb at the same rate as the primary tooth and be eliminated rapidly if accidentally extruded through the apex and have the ability for disinfection of pulpal and periapical lesion.

In this study 2 medications will be used as root canal filling. First is the mixture of zinc oxide eugenol based sealer (ZicalR) and 3mixtatin which is composed of 3 antibiotics (ciprofloxacin, cefixime, metronidazole), simvastatin, and zinc oxide the term 3mix-tatin as an acronym for the mixture of triple mixture antibiotics and simvastatin. Statin components are emerging material in regenerative endodontics. Clinical and experimental trials proved the pleiotropic effect of statin, as it increases the osteoblastic function and suppresses the osteoclastic function. In addition to that, evidence proved that it is a potent anti -inflammatory as it reduce the CRP and pro-inflammatory cytokines. Second medication will be Zical which is a zinc oxide eugenol based sealer composed of Zinc Oxide, Bismuth Sub-carbonate, Barium Sulphate, Sodium Borate, Iodoform, and Hydrogenated Resin. Liquid contains: Eugenol.

ELIGIBILITY:
Inclusion Criteria

1. Children age range from 5-7 years.
2. Children free from any systemic diseases or genetic disorders.
3. Primary molar with necrotic pulp, with pain, gingival abscess, sinus openings.
4. Clinical mobility not exceeding grade two.
5. Radiographic evidence of non-perforating internal resorption, external resorption not exceeding 1\3 of the root
6. Furcation or periapical radiolucency.

Exclusion Criteria:

1. Non-restorable molars or beyond repair, for example: decay reaches to bifurcation, a hard gingival margin cannot be established or infection cannot be eradicated by other mean (Balaji, 2007).
2. Patient with known allergy to any type of antibiotics or anti-hyperlipidemia drugs.
3. Patient with facial cellulitis or lymphadenopathy
4. Lack of patient/parent compliance and cooperation.
5. Refusal of participation or failure to obtain an informed consent.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | first week after treatment, 3 months, 6 months, 12 months
  spontaneous pain, as reported by the caregivers through visual analogue score (VAS)from 1 to 10 where 1 means : minimal pain , 10 means:: severe pain

SECONDARY OUTCOMES:
Root resorption | preoperative, 3rd month, 6 month, 12 month
  Presence of Radiographic internal or external root resorption in periapical radiograph using parallel technique
Bone resorption | preoperative, 3 , 6 , 12 month
  Presence of Radiographic bone resorption in periapical radiograph technique of Radiograph: extension cone paralelling periapical radiograph (XCP)

CONTACTS AND LOCATIONS:
Overall Officials: amira badran, Phd, Study Director — associate professor
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No